CLINICAL TRIAL: NCT00413322
Title: A Phase I Safety, Pharmacodynamic, Anti-Tumor Activity, and Pharmacokinetic Study of PXD101 Alone and in Combination With 5-Fluorouracil in Patients With Advanced Solid Tumors
Brief Title: Study of PXD101 Alone and in Combination With 5-Fluorouracil (5-FU) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-4
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Tumor
Keywords: Advanced Solid tumor; Adenosarcoma; Androgen-independent prostate cancer; belinostat; bladder cancer; bladder neoplasms; Breast cancer; Carcinoma, Bronchogenic; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Carcinosarcoma; Chondrosarcoma; Coin Lesion, Pulmonary; colorectal cancer; Esophageal Neoplasms; Facial Neoplasms; Fibrosarcoma; head and neck cancer; Hemangiosarcoma; Histiocytoma, Malignant Fibrous; kidney cancer; Leiomyosarcoma; Liposarcoma; lung cancer; lung neoplasms; Lymphangiosarcoma; mesothelioma; mesothelioma, cystic; Mixed Tumor, Mesodermal; Mouth Neoplasms; Myosarcoma; Myxosarcoma; Osteosarcoma; Otorhinolaryngologic Neoplasms; Ovarian cancer; Pancoast's Syndrome; Parathyroid Neoplasms; Phyllodes Tumor; Pulmonary Sclerosing Hemangioma; sarcoma; thyroid cancer; Thyroid Neoplasms; Tracheal Neoplasms; PXD101
MeSH Terms: conditions — Neoplasms; Adenosarcoma; Urinary Bladder Neoplasms; Breast Neoplasms; Carcinoma, Bronchogenic; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Carcinosarcoma; Chondrosarcoma; Solitary Pulmonary Nodule; Colorectal Neoplasms; Esophageal Neoplasms; Facial Neoplasms; Fibrosarcoma; Head and Neck Neoplasms; Hemangiosarcoma; Histiocytoma, Malignant Fibrous; Kidney Neoplasms; Leiomyosarcoma; Liposarcoma; Lung Neoplasms; Lymphangiosarcoma; Mesothelioma; Mesothelioma, Cystic; Mixed Tumor, Mesodermal; Mouth Neoplasms; Myosarcoma; Myxosarcoma; Osteosarcoma; Otorhinolaryngologic Neoplasms; Ovarian Neoplasms; Pancoast Syndrome; Parathyroid Neoplasms; Phyllodes Tumor; Pulmonary Sclerosing Hemangioma; Sarcoma; Thyroid Neoplasms; Tracheal Neoplasms | interventions — belinostat; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm dose escalation (Experimental)
  Interventions: Drug: belinostat; Drug: 5-Fluorouracil (5-FU)

INTERVENTIONS:
Drug: belinostat — 300, 600, or 1000 mg/m2 belinostat IV for 5 days every 21 days starting with cycle 1
  Other Names: PXD101
Drug: 5-Fluorouracil (5-FU) — 250, 500, 750, or 1000 mg/m2/d of 5-FU starting with cycle 2 onwards in combination with belinostat. Starting on day 2, 5-FU is administered as a continuous 96 hour infusion.
  Other Names: 5-FU

SUMMARY:
This is a study to assess the combination of PXD101 and 5-Fluorouracil (5-FU)in patients with advanced solid tumors. The primary goal of the study is to understand the safety, anti-tumor activity, and how the study drug behaves within the body when given with 5-Fluorouracil (5-FU).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors
* Advanced colorectal cancer or other adenocarcinomas
* Tumor progression after standard chemotherapy, or where none yet approved
* At least one unidimensionally measurable lesion
* Karnofsky performance >= 70%
* Life expectancy of at least 3 months
* Age >= 18 years
* Signed, written Institutional Review Board (IRB)-approved informed consent
* Acceptable liver function:

  * Bilirubin <= 1.5 x upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) <= 2.5 x ULN, OR
  * AST (SGOT) and ALT (SGPT) <= 5 x ULN if liver metastasis
* Acceptable renal function:

  * Serum creatinine within normal limits, OR
  * Calculated creatinine clearance of >= 60 mL/min/1.73 m2 for certain patients
* Acceptable hematologic status:

  * Absolute neutrophil count (ANC) >= 1500 cells/mm3
  * Platelet count >= 100,000 (plt/mm3)
  * Hemoglobin >= 9 g/dL
* Urinalysis: No clinically significant abnormalities
* Acceptable coagulation status:

  * Prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits, OR
  * For patients on anticoagulation therapy, status within therapeutic range
* For men and women of child-producing potential, use of effective contraception
* Tumors accessible for needle biopsy

Exclusion Criteria:

* Significant cardiovascular disease.
* A marked baseline prolongation of QT/QTc interval
* Long QT syndrome
* Required use of medication on dosing days that may cause torsade de pointes.
* Infections requiring intravenous (IV) systemic therapy
* Pregnant or nursing women
* Treatment with chemotherapy or investigational therapy < 4 weeks (28 days) prior to study entry (6 weeks for nitrosoureas, mitomycin C, or Avastin).
* Treatment with radiation therapy or surgery either within 2 weeks prior to study entry, or not yet recovered if 2-4 weeks prior to study entry.
* Unwillingness or inability to comply with protocol procedures.
* Known active uncontrolled infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease (e.g. hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Concurrent use of other investigational agent(s)
* Serious concurrent medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
to determine the maximum tolerated dose of PXD101 administered in combination with 5-FU | throughout the study
to determine whether PXD101 alone can down-regulate thymidylate synthase in patient tumors | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Topotarget A/S, Study Chair — Valerio Therapeutics
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Nebraska, Omaha, Nebraska
  - Portsmouth Regional Hospital Hematology/Oncology Clinic, Portsmouth, New Hampshire